CLINICAL TRIAL: NCT05437484
Title: Design, Implementation and Evaluation of a Peer-led Alcohol Prevention Intervention for College Students. A Exploratory Trial
Brief Title: Peer-led Brief Alcohol Intervention for College Student Drinkers in Spain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Sara Pueyo, Clinical nurse, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SP EXPLORATORIO
Record Dates: First submitted 2022-06-16; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Peer Group; Motivational Interviewing; Cognitive Behavioral Therapy; Alcohol Drinking in College
Keywords: Brief interventions; Motivational interviewing; Peer counsellors; College students; Alcohol; Counsellor behavior
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: peer-led BASICS session (Experimental): Participants randomized to the intervention group received a peer-led BASICS session.
  Interventions: Behavioral: Peer-led BASICS
- Control group (No Intervention): Participants randomized to the control group did not receive any specific intervention.

INTERVENTIONS:
Behavioral: Peer-led BASICS — The peer-led BASICS session consisted in a face-to-face 50-minute motivational interview. In this meeting, the peer counsellor oriented the participant using a personalized graphic feedback sheet, with topics including participant's drinking pattern; level of intoxication; perceived and actual descriptive drinking norms, alcohol expectancies; drinking consequences; individual risk factors; financial costs; alcohol caloric consumption, and hours of exercise required to burn those calories, and protective behavioral strategies. Participants received a copy of the personalized feedback, a personalized BAC card, and a tips sheet.
  BASICS facilitators were volunteer undergraduate nursing students from who attented a pre-training course and showed being competent to conduct BASICS-based motivational interview and knowledgeable about alcohol.
  Arms: Intervention group: peer-led BASICS session

SUMMARY:
A pilot randomized controlled trial was carried out. Fifty nursing students were randomly assigned either a 50-minute brief motivational intervention with individual feedback or a treatment-as-usual control condition. The intervention was delivered by undergraduate peer counsellors trained in Brief Alcohol Screening and Intervention for College Students. Primary outcomes for testing efficacy were alcohol use and alcohol-related consequences.

DETAILED DESCRIPTION:
Aims: To assess the potential efficacy and the feasibility of a peer-led brief alcohol intervention aimed to reduce the alcohol consumption in Spanish heavy nursing student drinkers.

Methods: A pilot randomized controlled trial was carried out. Fifty nursing students were randomly assigned either a 50-minute brief motivational enhancement intervention with individual feedback (n=23) or a treatment-as-usual control condition (n=27). Both motivational interviewing and personalized feedback were delivered by undergraduate peer counsellors trained in Brief Alcohol Screening and Intervention for College Students (BASICS). Participants were assessed during their pledge year of university with a one-month follow-up. Primary outcomes for testing efficacy were alcohol use (quantity, heavy-drinking episodes, and peak blood alcohol concentration), and alcohol-related consequences. Quantitative data were analyzed using the U-Mann-Whitney and Wilcoxon test. Content analysis was used for measuring the feasibility of the program.

ELIGIBILITY:
Inclusion Criteria:

* First year university students of Nursing Degree, between 18 and 20 years old.
* Students of first access to the University.
* Having had at least one episode of heavy drinking or binge drinking in the past month.

Exclusion Criteria:

* Students who have started or previously studied other university degrees or a higher degree.
* University students who do not consume alcohol or, if they do consume alcohol, have not had binge drinking in the last month.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in 'Quantitaty of alcohol use in a typical weekend' (preliminary efficacy outcomes) | For measuring the change, there are two time points: pre-test and post-test (one month after receiving the programme)
  Assesing the change in the total number of drinks during a typical weekend (Thursday, Friday, Saturday and Sunday) during the previous 30 days.
Change in 'Estimated peak blood alcohol content (peak BAC)' (preliminary efficacy outcomes) | For measuring the change, there are two time points: pre-test and post-test (one month after receiving the programme)
  Assesing the change in the estimated peak blood alcohol content. It was calculated using participants' responses about maximum drinks consumed on the occasion of highest consumption in the last month, and the number of hours they spent drinking on that occasion.
Change in 'Frequency of binge drinking episodes' (preliminary efficacy outcomes) | For measuring the change, there are two time points: pre-test and post-test (one month after receiving the programme)
  Assesing the change in the frequency of binge drinking episodes in the past month (5 or more (male)/ 4 or more (female) glasses of alcoholic beverages on the same drinking occasion).
Change in 'Number of alcohol-related consequences (preliminary efficacy outcomes)' | For measuring the change, there are two time points: pre-test and post-test (one month after receiving the programme)
  Assesing the change in the number of negative consequences associated with their alcohol consumption in the previous 30 days.

SECONDARY OUTCOMES:
Peer counselors' fidelity -adherence to motivational interviewing skills and alcohol-related content (feasibility outcomes) | From the beginning of the intervention sessions until the end of the intervention, an average of 3 months.
  Peer counselors' fidelity to the implementation of the intervention, including adherence to the theoretical alchol-related content, and the use of MI skills during the intervention.
  For their measurement, an alcohol-related content checklist and the Peer Proficiency Assessment were used.
Barriers and facilitators of the implementation process (feasibility outcomes) | From the beginning of the peer counsellors' training until the end of the intervention, an average of 9 months.
  Factors that have affected positively and negatively during the program implementation.
Acceptability -satisfaction- (feasibility outcomes) | From the beginning of the intervention sessions until the end of the intervention, an average of 3 months.
  Satisfaction of both participants and peer counsellors with the program. It was used and ad-hoc questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No